CLINICAL TRIAL: NCT02922062
Title: The Effects of Palm Oil Consumed Under Different Macronutrient Distributions on Circulating Lipoprotein and Fatty Acid Profiles
Brief Title: The Effects of Consuming Palm Oil With Different Macronutrient Intakes on Blood Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Malaysia Palm Oil Board (Other Government)
Responsible Party: Principal Investigator, Jeff Volek, Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GRT00038995
Record Dates: First submitted 2016-06-17; First posted 2016-10-03 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Cardiovascular Diseases; Inflammation
Keywords: lipids; saturated fat; palm oil
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Rapeseed Oil; Palm Oil; Fatty Acids; Butter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Carbohydrate Diet (Experimental): Half of the participants will be randomly assigned to this diet arm. The macronutrient composition of the diet will be (PRO (protein):CHO (carbohydrate):FAT, 18:8:74). There are three diet phases within this arm that use different fats as the primary cooking oil either canola oil, palm oil or butter. Each diet phase lasts for 3 weeks. At the end of each diet phase the testing battery completed at baseline will be repeated followed by a 2 week washout where subjects revert back to their usual diets. Canola oil is the low saturated fat control diet and is administered first. Participants then randomly begin either the palm oil or canola oil diet phases.
  Interventions: Other: Canola Oil; Other: Palm Oil; Other: Butter
- High Carbohydrate Diet (Active Comparator): Half of the participants will be randomly assigned to this diet arm. The macronutrient composition of the diet will be (PRO:CHO:FAT, 18:60:22). There are three diet phases within this arm that use different fats as the primary cooking oil either canola oil, palm oil or butter. Each diet phase lasts for 3 weeks. At the end of each diet phase the testing battery completed at baseline will be repeated followed by a 2 week washout where subjects revert back to their usual diets. Canola oil is the low saturated fat control diet and is administered first. Participants then randomly begin either the palm oil or canola oil diet phases.
  Interventions: Other: Canola Oil; Other: Palm Oil; Other: Butter

INTERVENTIONS:
Other: Canola Oil — Subjects will be provided with all their meals prepared in our metabolic kitchen in order to control their diets. The major cooking oil used in food preparation will be canola oil. The meals will be tailored to the caloric needs of each individual in order to maintain their body weight.
  Other Names: low saturated fat control; Controlled Dietary Intervention using Canola Oil
Other: Palm Oil — Subjects will be provided with all their meals prepared in our metabolic kitchen in order to control their diets. The major cooking oil used in food preparation will be palm oil. The meals will be tailored to the caloric needs of each individual in order to maintain their body weight.
  Other Names: saturated fat; Controlled Dietary Intervention using Palm Oil
Other: Butter — Subjects will be provided with all their meals prepared in our metabolic kitchen in order to control their diets. The major cooking oils used in food preparation will be butter. The meals will be tailored to the caloric needs of each individual in order to maintain their body weight.
  Other Names: saturated fat; Controlled Dietary Intervention using Butter

SUMMARY:
The purpose of this study is to determine the effects of palm oil when consumed as either part of a low carbohydrate diet or a high carbohydrate diet on blood lipids, cardiovascular health and inflammation. The study will help us better understand how the quality of saturated fat and the quantity of carbohydrate interact to impact blood lipids and cardiovascular health.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of palm oil on blood lipids, cardiovascular health and inflammation. Potential subjects will be screened until 24 qualifying healthy participants are enrolled. After enrollment participants will undergo a baseline battery of tests including blood draws, body composition, measures of height and weight, blood lipid profile (cholesterol, lipoprotein particle size, quantity and fatty acid composition), insulin sensitivity using a static index, inflammation, antioxidant status and measurement of energy expenditure and substrate oxidation by indirect calorimetry. Participants will be randomly divided into one of two arms/tracks, either a low carbohydrate diet arm or a high carbohydrate diet arm. Each diet arm consists of 3 phases a low saturated fat control diet where the primary cooking oil is canola oil and two saturated fat diet phases where the primary cooking oil is either palm oil or butter.

Participants will begin with the low saturated fat diet phase first which consists of 50% of fat calories derived from canola oil for 3 weeks. At the end of this control diet phase the battery of tests completed at baseline will be repeated. After a 2-week washout period participants will then proceed in random order into either the palm oil or butter diet phases of their diet arm/track. The palm oil and butter diet phases are also 3 weeks in duration and separated by a 2 week washout period. The palm oil and butter diet phases will derive 50% of the fat calories from either palm oil or butter. Both oils are high in saturated fat but differ in the quality of saturated fat. At the end of each diet phase the testing battery completed at baseline will be repeated. The subjects will never be exposed to more than minimal risk and in return will receive 9 weeks of food, individualized reports of their study results and a monetary stipend. The study will help us better understand how the quality of saturated fat and the quantity of carbohydrate interact to impact blood lipids and cardiovascular health. This knowledge can be used to aid dietary recommendations for cardiovascular health and control of blood lipids.

ELIGIBILITY:
Inclusion Criteria:

* normocholesterolemic

Exclusion Criteria:

* hypercholesterolemia
* diabetes
* liver disease
* kidney disease
* other metabolic or endocrine dysfunction
* diagnosis of cancer within the previous 5 years
* hypertension
* current use of cholesterol reducing medications
* current use of diabetic medications

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in High-Density Lipoprotein (HDL) Particle Size between Canola Oil and Palm Oil Diet Phases (Part of the Lipoprotein Distribution) | Assessed during the 3rd week of the canola oil and palm oil diet
  The change in HDL particle size and the number of each size particle between Canola Oil and Palm Oil diets will be assessed by Nuclear Magnetic Resonance (NMR) spectroscopy
Change in HDL Particle Size between Canola Oil and Butter Diet Phases (Part of the Lipoprotein Distribution) | Assessed during the 3rd week of the canola oil and butter diets
  The change in HDL particle size and the number of each size particle between Canola Oil and Butter diets will be assessed by Nuclear Magnetic Resonance (NMR) spectroscopy
Change in Low-Density Lipoprotein (LDL) Particle Size between Canola Oil and Palm Oil Diet Phases (Part of the Lipoprotein Distribution) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in LDL particle size and the number of each size particle between Canola Oil and Palm Oil diets will be assessed by NMR spectroscopy
Change in LDL Particle Size between Canola Oil and Butter Diet Phases (Part of the Lipoprotein Distribution) | Assessed during the 3rd week of the canola oil and butter diets
  The change in LDL particle size and the number of each size particle between Canola Oil and Palm Oil diets will be assessed by NMR spectroscopy
Change in Very Low-Density Lipoprotein (VLDL) Particle Size between Canola Oil and Palm Oil Diet Phases (Part of the Lipoprotein Distribution) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in VLDL particle size and the number of each size particle between Canola Oil and Palm Oil diets will be assessed by NMR spectroscopy
Change in VLDL Particle Size between Canola Oil and Butter Diet Phases (Part of the Lipoprotein Distribution) | Assessed during the 3rd week of the canola oil and butter diets
  The change in VLDL particle size and the number of each size particle between Canola and Butter diets will be assessed by NMR spectroscopy

SECONDARY OUTCOMES:
Change in Insulin Sensitivity between the Canola Oil and Palm Oil Diet Phases | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in glucose and insulin between Canola Oil and Palm Oil diets will be measured from plasma to determine the Homeostasis Model Assessment (HOMA) index score
Change in Insulin Sensitivity between the Canola Oil and Butter Diet Phases | Assessed during the 3rd week of the canola oil and butter diets
  The change in glucose and insulin between Canola Oil and Palm Oil diets will be measured from plasma to determine the Homeostasis Model Assessment (HOMA) index score
Change in Body Weight between the Canola Oil and Palm Oil Diet Phases | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in body mass between Canola Oil and Palm Oil diets will be measured on a scale
Change in Body Weight between the Canola Oil and Butter Diet Phases | Assessed during the 3rd week of the canola oil and butter diets
  The change in body mass between Canola Oil and Butter diets will be measured on a scale
Change in Body Composition (Percent of Lean Mass, Fat Mass and Bone Mass according to the 3-compartment Model) between the Canola Oil and Palm Oil Diet Phases | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in body composition between Canola Oil and Palm Oil diets will be measured by dual-energy X-ray absorptiometry
Change in Body Composition (Percent of Lean Mass, Fat Mass and Bone Mass according to the 3-compartment Model) between the Canola Oil and Butter Diet Phases | Assessed during the 3rd week of the canola oil and butter diets
  The change in body composition between Canola Oil and Butter diets will be measured by dual-energy X-ray absorptiometry
Change in the Cholesterol Profile between the Canola Oil and Palm Oil Diet Phases (Part of the Cholesterol Profile) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in total cholesterol and HDL cholesterol between Canola Oil and Palm Oil diets will be measured by immunoturbidimetry and LDL cholesterol will be calculated using these two values.
Change in the Cholesterol Profile between the Canola Oil and Butter Diet Phases (Part of the Cholesterol Profile) | Assessed during the 3rd week of the canola oil and butter diets
  The change in total cholesterol and HDL cholesterol between Canola Oil and Butter diets will be measured by immunoturbidimetry and LDL cholesterol will be calculated using these two values.
Change in Total Triglycerides between the Canola Oil and Palm Oil Diet Phases (Part of the Cholesterol Profile) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in triglycerides between Canola Oil and Palm Oil diets will be measured by immunoturbidimetry
Change in Total Triglycerides between the Canola Oil and Butter Diet Phases (Part of the Cholesterol Profile) | Assessed during the 3rd week of the canola oil and butter diets
  The change in triglycerides between Canola Oil and Butter diets will be measured by immunoturbidimetry
Change in the Apolopoprotein-A1 Concentration in plasma between the Canola Oil and Palm Oil Diet Phases (Part of the Cholesterol Profile) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in Apolopoprotein-A1 between Canola Oil and Palm Oil diets will be assessed by ELISA
Change in the Apolopoprotein-A1 Concentration in plasma between the Canola Oil and Butter Diet Phases (Part of the Cholesterol Profile) | Assessed during the 3rd week of the canola oil and butter diets
  The change in Apolopoprotein-A1 between Canola Oil and Butter diets will be assessed by ELISA
Change in the Apolopoprotein-B Concentration in plasma between the Canola Oil and Palm Oil Diet Phases (Part of the Cholesterol Profile) | Assessed during the 3rd week of the canola oil and Palm Oil diets
  The change in Apolopoprotein-B between Canola Oil and Palm Oil diets will be assessed by ELISA
Change in the Apolopoprotein-B Concentration in plasma between the Canola Oil and Butter Diet Phases (Part of the Cholesterol Profile) | Assessed during the 3rd week of the canola oil and butter diets
  The change in Apolopoprotein-B between Canola Oil and Butter Diets will be assessed by ELISA
Change in the Fatty Acid Composition of the Plasma between the Canola Oil and Palm Oil Diet Phases | Assessed during the 3rd week of the canola oil and palm oil diets
  Teh change in the fatty acid composition of the plasma between Canola Oil and Palm Oil diets will be assessed by gas chromatography using flame ionization detection
Change in the Fatty Acid Composition of the Plasma between the Canola Oil and Butter Diet Phases | Assessed during the 3rd week of the canola oil and butter diets
  The change in the fatty acid composition of the plasma between Canola Oil and Butter will be assessed by gas chromatography using flame ionization detection

OTHER OUTCOMES:
Change in C-Reactive Protein between the Canola Oil and Palm Oil Diet Phases (Part of an Inflammatory Panel) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in C-Reactive Protein between Canola Oil and Palm Oil diets will be assessed using a multiplex ELISA platform
Change in C-Reactive Protein between the Canola Oil and Butter Diet Phases (Part of an Inflammatory Panel) | Assessed during the 3rd week of the canola oil and butter diets
  The change in C-Reactive Protein between Canola Oil and Palm Oil diets will be assessed using a multiplex ELISA platform
Change in Interleukin (IL)-1beta Protein between the Canola Oil and Palm Oil Diet Phases (Part of an Inflammatory Panel) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in IL-1beta between Canola Oil and Palm Oil diets will be assessed using a multiplex ELISA platform
Change in IL-1beta Protein between the Canola Oil and Butter Diet Phases (Part of an Inflammatory Panel) | Assessed during the 3rd week of the canola oil and butter diets
  The change in IL-1beta between Canola Oil and Butter diets will be assessed using a multiplex ELISA platform
Change in Tumor Necrosis Factor (TNF)-alpha between the Canola Oil and Palm Oil Diet Phases (Part of an Inflammatory Panel) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in TNF-alpha between Canola Oil and Palm Oil diets will be assessed using a multiplex ELISA platform
Change in TNF-alpha between the Canola Oil and Butter Diet Phases (Part of an Inflammatory Panel) | Assessed during the 3rd week of the canola oil and butter diets
  The change in TNF-alpha between Canola Oil and Palm Oil will be assessed using a multiplex ELISA platform
Change in Neopterin between the Canola Oil and Palm Oil Diet Phases (Part of an Inflammatory Panel) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in TNF-alpha between Canola Oil and Palm Oil diets will be assessed using a singleplex ELISA platform
Change in Neopterin between the Canola Oil and Butter Diet Phases (Part of an Inflammatory Panel) | Assessed during the 3rd week of the canola oil and butter diets
  The change in Neopterin between Canola Oil and Butter diets will be assessed using a singleplex ELISA platform
Change in Elastase between the Canola Oil and Palm Oil Diet Phases (Part of an Inflammatory Panel) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in Elastase between Canola Oil and Palm Oil diets will be assessed using a singleplex ELISA platform
Change in Elastase between the Canola Oil and Butter Diet Phases (Part of an Inflammatory Panel) | Assessed during the 3rd week of the canola oil and butter diets
  The change in Elastase between Canola Oil and Butter diets will be assessed using a singleplex ELISA platform
Change in Conjugated Dienes between the Canola Oil and Palm Oil Diet Phases (Part of an Antioxidant Status Assessment) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in Conjugated dienes, an early stage lipid peroxidation product, between Canola Oil and Palm Oil diets will be assessed by spectrophotometry.
Change in Conjugated Dienes between the Canola Oil and Butter Diet Phases (Part of an Antioxidant Status Assessment) | Assessed during the 3rd week of the canola oil and butter diets
  The change in Conjugated dienes, an early stage lipid peroxidation product, between Canola Oil and Butter diets will be assessed by spectrophotometry.
Change in Malondialdehyde between the Canola Oil and Palm Oil Diet Phases (Part of an Antioxidant Status Assessment) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in Malondialdehyde, a late stage lipid peroxidation product, between Canola Oil and Palm Oil diets will be assessed by spectroscopy.
Change in Malondialdehyde between the Canola Oil and Butter Diet Phases (Part of an Antioxidant Status Assessment) | Assessed during the 3rd week of the canola oil and butter diets
  The change in Malondialdehyde, a late stage lipid peroxidation product, between Canola Oil and Butter diets will be assessed by high performance liquid chromatography.
Change in the Total Antioxidant Capacity of the blood between the Canola Oil and Palm Oil Diet Phases (Part of an Antioxidant Status Assessment) | Assessed during the 3rd week of the canola oil and palm oil diets
  The change in the total antioxidant capacity of the blood between Canola Oil and Palm Oil diets will be assessed by spectrophotometry using the Ferric Reducing Antioxidant Power (FRAP) assay.
Change in the Total Antioxidant Capacity of the blood between the Canola Oil and Butter Diet Phases (Part of an Antioxidant Status Assessment) | Assessed during the 3rd week of the canola oil and butter diets
  The change in the total antioxidant capacity of the blood between Canola Oil and Butter diets will be assessed by spectrophotometry using the FRAP assay.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Volek, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- Physical Activity and Education Services (PAES) Building, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with other scientists but participants will be provided with their own individual data when the study is complete.

REFERENCES:
- [Background] Clarke R, Frost C, Collins R, Appleby P, Peto R. Dietary lipids and blood cholesterol: quantitative meta-analysis of metabolic ward studies. BMJ. 1997 Jan 11;314(7074):112-7. doi: 10.1136/bmj.314.7074.112. PMID 9006469
- [Background] de Lorgeril M, Salen P, Martin JL, Monjaud I, Delaye J, Mamelle N. Mediterranean diet, traditional risk factors, and the rate of cardiovascular complications after myocardial infarction: final report of the Lyon Diet Heart Study. Circulation. 1999 Feb 16;99(6):779-85. doi: 10.1161/01.cir.99.6.779. PMID 9989963
- [Background] Howard BV, Van Horn L, Hsia J, Manson JE, Stefanick ML, Wassertheil-Smoller S, Kuller LH, LaCroix AZ, Langer RD, Lasser NL, Lewis CE, Limacher MC, Margolis KL, Mysiw WJ, Ockene JK, Parker LM, Perri MG, Phillips L, Prentice RL, Robbins J, Rossouw JE, Sarto GE, Schatz IJ, Snetselaar LG, Stevens VJ, Tinker LF, Trevisan M, Vitolins MZ, Anderson GL, Assaf AR, Bassford T, Beresford SA, Black HR, Brunner RL, Brzyski RG, Caan B, Chlebowski RT, Gass M, Granek I, Greenland P, Hays J, Heber D, Heiss G, Hendrix SL, Hubbell FA, Johnson KC, Kotchen JM. Low-fat dietary pattern and risk of cardiovascular disease: the Women's Health Initiative Randomized Controlled Dietary Modification Trial. JAMA. 2006 Feb 8;295(6):655-66. doi: 10.1001/jama.295.6.655. PMID 16467234
- [Background] Krauss RM. Lipoprotein subfractions and cardiovascular disease risk. Curr Opin Lipidol. 2010 Aug;21(4):305-11. doi: 10.1097/MOL.0b013e32833b7756. PMID 20531184
- [Background] Cromwell WC, Otvos JD, Keyes MJ, Pencina MJ, Sullivan L, Vasan RS, Wilson PW, D'Agostino RB. LDL Particle Number and Risk of Future Cardiovascular Disease in the Framingham Offspring Study - Implications for LDL Management. J Clin Lipidol. 2007 Dec;1(6):583-92. doi: 10.1016/j.jacl.2007.10.001. PMID 19657464
- [Background] Warensjo E, Riserus U, Vessby B. Fatty acid composition of serum lipids predicts the development of the metabolic syndrome in men. Diabetologia. 2005 Oct;48(10):1999-2005. doi: 10.1007/s00125-005-1897-x. Epub 2005 Aug 13. PMID 16132958
- [Background] Zong G, Zhu J, Sun L, Ye X, Lu L, Jin Q, Zheng H, Yu Z, Zhu Z, Li H, Sun Q, Lin X. Associations of erythrocyte fatty acids in the de novo lipogenesis pathway with risk of metabolic syndrome in a cohort study of middle-aged and older Chinese. Am J Clin Nutr. 2013 Aug;98(2):319-26. doi: 10.3945/ajcn.113.061218. Epub 2013 Jun 26. PMID 23803879
- [Background] Hodge AM, English DR, O'Dea K, Sinclair AJ, Makrides M, Gibson RA, Giles GG. Plasma phospholipid and dietary fatty acids as predictors of type 2 diabetes: interpreting the role of linoleic acid. Am J Clin Nutr. 2007 Jul;86(1):189-97. doi: 10.1093/ajcn/86.1.189. PMID 17616780
- [Background] Wang L, Folsom AR, Zheng ZJ, Pankow JS, Eckfeldt JH; ARIC Study Investigators. Plasma fatty acid composition and incidence of diabetes in middle-aged adults: the Atherosclerosis Risk in Communities (ARIC) Study. Am J Clin Nutr. 2003 Jul;78(1):91-8. doi: 10.1093/ajcn/78.1.91. PMID 12816776
- [Background] Kroger J, Zietemann V, Enzenbach C, Weikert C, Jansen EH, Doring F, Joost HG, Boeing H, Schulze MB. Erythrocyte membrane phospholipid fatty acids, desaturase activity, and dietary fatty acids in relation to risk of type 2 diabetes in the European Prospective Investigation into Cancer and Nutrition (EPIC)-Potsdam Study. Am J Clin Nutr. 2011 Jan;93(1):127-42. doi: 10.3945/ajcn.110.005447. Epub 2010 Oct 27. PMID 20980488
- [Background] Patel PS, Sharp SJ, Jansen E, Luben RN, Khaw KT, Wareham NJ, Forouhi NG. Fatty acids measured in plasma and erythrocyte-membrane phospholipids and derived by food-frequency questionnaire and the risk of new-onset type 2 diabetes: a pilot study in the European Prospective Investigation into Cancer and Nutrition (EPIC)-Norfolk cohort. Am J Clin Nutr. 2010 Nov;92(5):1214-22. doi: 10.3945/ajcn.2010.29182. Epub 2010 Sep 22. PMID 20861175
- [Background] Vessby B, Aro A, Skarfors E, Berglund L, Salminen I, Lithell H. The risk to develop NIDDM is related to the fatty acid composition of the serum cholesterol esters. Diabetes. 1994 Nov;43(11):1353-7. doi: 10.2337/diab.43.11.1353. PMID 7926311
- [Background] Mahendran Y, Agren J, Uusitupa M, Cederberg H, Vangipurapu J, Stancakova A, Schwab U, Kuusisto J, Laakso M. Association of erythrocyte membrane fatty acids with changes in glycemia and risk of type 2 diabetes. Am J Clin Nutr. 2014 Jan;99(1):79-85. doi: 10.3945/ajcn.113.069740. Epub 2013 Oct 23. PMID 24153340
- [Background] Miettinen TA, Naukkarinen V, Huttunen JK, Mattila S, Kumlin T. Fatty-acid composition of serum lipids predicts myocardial infarction. Br Med J (Clin Res Ed). 1982 Oct 9;285(6347):993-6. doi: 10.1136/bmj.285.6347.993. PMID 6812744
- [Background] Simon JA, Hodgkins ML, Browner WS, Neuhaus JM, Bernert JT Jr, Hulley SB. Serum fatty acids and the risk of coronary heart disease. Am J Epidemiol. 1995 Sep 1;142(5):469-76. doi: 10.1093/oxfordjournals.aje.a117662. PMID 7677125
- [Background] Wang L, Folsom AR, Eckfeldt JH. Plasma fatty acid composition and incidence of coronary heart disease in middle aged adults: the Atherosclerosis Risk in Communities (ARIC) Study. Nutr Metab Cardiovasc Dis. 2003 Oct;13(5):256-66. doi: 10.1016/s0939-4753(03)80029-7. PMID 14717057
- [Background] Yamagishi K, Nettleton JA, Folsom AR; ARIC Study Investigators. Plasma fatty acid composition and incident heart failure in middle-aged adults: the Atherosclerosis Risk in Communities (ARIC) Study. Am Heart J. 2008 Nov;156(5):965-74. doi: 10.1016/j.ahj.2008.06.017. Epub 2008 Aug 29. PMID 19061714
- [Background] Chowdhury R, Warnakula S, Kunutsor S, Crowe F, Ward HA, Johnson L, Franco OH, Butterworth AS, Forouhi NG, Thompson SG, Khaw KT, Mozaffarian D, Danesh J, Di Angelantonio E. Association of dietary, circulating, and supplement fatty acids with coronary risk: a systematic review and meta-analysis. Ann Intern Med. 2014 Mar 18;160(6):398-406. doi: 10.7326/M13-1788. PMID 24723079
- [Background] Chavarro JE, Kenfield SA, Stampfer MJ, Loda M, Campos H, Sesso HD, Ma J. Blood levels of saturated and monounsaturated fatty acids as markers of de novo lipogenesis and risk of prostate cancer. Am J Epidemiol. 2013 Oct 15;178(8):1246-55. doi: 10.1093/aje/kwt136. Epub 2013 Aug 28. PMID 23989197
- [Background] Forsythe CE, Phinney SD, Fernandez ML, Quann EE, Wood RJ, Bibus DM, Kraemer WJ, Feinman RD, Volek JS. Comparison of low fat and low carbohydrate diets on circulating fatty acid composition and markers of inflammation. Lipids. 2008 Jan;43(1):65-77. doi: 10.1007/s11745-007-3132-7. Epub 2007 Nov 29. PMID 18046594
- [Background] Forsythe CE, Phinney SD, Feinman RD, Volk BM, Freidenreich D, Quann E, Ballard K, Puglisi MJ, Maresh CM, Kraemer WJ, Bibus DM, Fernandez ML, Volek JS. Limited effect of dietary saturated fat on plasma saturated fat in the context of a low carbohydrate diet. Lipids. 2010 Oct;45(10):947-62. doi: 10.1007/s11745-010-3467-3. Epub 2010 Sep 7. PMID 20820932
- [Background] Volek JS, Phinney SD, Forsythe CE, Quann EE, Wood RJ, Puglisi MJ, Kraemer WJ, Bibus DM, Fernandez ML, Feinman RD. Carbohydrate restriction has a more favorable impact on the metabolic syndrome than a low fat diet. Lipids. 2009 Apr;44(4):297-309. doi: 10.1007/s11745-008-3274-2. Epub 2008 Dec 12. PMID 19082851
- [Background] Volk BM, Kunces LJ, Freidenreich DJ, Kupchak BR, Saenz C, Artistizabal JC, Fernandez ML, Bruno RS, Maresh CM, Kraemer WJ, Phinney SD, Volek JS. Effects of step-wise increases in dietary carbohydrate on circulating saturated Fatty acids and palmitoleic Acid in adults with metabolic syndrome. PLoS One. 2014 Nov 21;9(11):e113605. doi: 10.1371/journal.pone.0113605. eCollection 2014. PMID 25415333
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Otvos JD, Jeyarajah EJ, Bennett DW, Krauss RM. Development of a proton nuclear magnetic resonance spectroscopic method for determining plasma lipoprotein concentrations and subspecies distributions from a single, rapid measurement. Clin Chem. 1992 Sep;38(9):1632-8. PMID 1326420